CLINICAL TRIAL: NCT04147065
Title: Helicobacter Pylori Eradication According to DPO-PCR Methods: Duration of Triple Therapy and Bismuth Quadruple According to Clarithromycin Resistance Patterns (K-CREATE Study)
Brief Title: Helicobacter Pylori Eradication According to DPO-PCR Methods (K-CREATE) Study)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Joon Sung Kim, Assistant professor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Incheon HP
Record Dates: First submitted 2019-10-20; First posted 2019-10-31 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter; Empirical; Tailored
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Phase I study Tailored therapy (Clar S: 7 vs. 14 d triple therapy, Clar R: 7 vs. 14d BQT) vs. empirical therapy (7 or 14 d triple therapy) for H. pylori eradication
  Phase 2 study Tailored therapy (Clar S: 7d triple therapy, Clar R: 7d BQT vs. empirical therapy (14d triple therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-day triple therapy and 7-day bismuth quadruple therapy (Experimental): 7-day triple therapy is consisted of proton pump inhibitor (PPI), amoxicillin and clarithromycin for seven days 7-day bismuth quadruple therapy is consisted of PPI, bismuth, tetracycline, metronidazole for seven days
  Interventions: Drug: Duration of eradication regimen
- 14-day triple therapy and 14-day bismuth quadruple therapy (Active Comparator): 14-day triple therapy is consisted of PPI, amoxicillin and clarithromycin for fourteen days 14-day bismuth quadruple therapy is consisted of PPI, bismuth, tetracycline, metronidazole for fourteen days
  Interventions: Drug: Duration of eradication regimen

INTERVENTIONS:
Drug: Duration of eradication regimen — 14 day eradication regimen
  Other Names: 14 day treatment

SUMMARY:
Clarithromycin-containing triple therapy is still the primary therapy approved by the Korean government. However, studies of antibiotic resistance have shown that regional resistance patterns to antibiotics such as clarithromycin are increasing. Recent studies show that examining genotype resistance is effective in eradication. Currently, dual priming oligonucleotide-polymerase chain reaction (DPO-PCR) is used to measure clarithromycin resistance. No study has compared the duration of eradication regimens according to DPO-PCR results. This study compares the eradication rate of 7-day triple therapy with 14-day triple therapy in clarithromycin susceptible strains from DPO-PCR. The investigators also aimed to compare the eradication rates of 7-day bismuth quadruple therapy with 14-day bismuth quadruple therapy from clarithromycin-resistant strains from DPO-PCR.

DETAILED DESCRIPTION:
This is a multi-center study performed at 20 university hospitals. The study is composed of two phases. In phase I, patients with H. pylori infection are randomized to receive tailored or empirical therapy. The empirical therapy group is further randomized to receive either 7-day triple therapy or 14-day triple therapy. The tailored group is randomized to receive triple therapy if they are clarithromycin sensitive or bismuth quadruple therapy if they are clarithromycin resistant. Each group is further randomized to receive either seven or 14 days of treatment. The eradication rates and adverse events of each regimen will be investigated.

In phase 2, patients with H. pylori infection are randomized to receive tailored or empirial therapy. The empirical therapy group receives 14 days of triple therapy. The tailored therapy group receives 7-day triple therapy if they are clarithromycin sensitive and 7-day bismuth quadruple therapy if clarithromycin resistant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had upper endoscopic examination within 3 months and diagnosed by Helicobacter pylori infection either by rapid urease test, urea breath test, or histopathologic examination.

Participants who voluntarily want to participate in this study.

Exclusion Criteria:

History of H. pylori eradication History of stomach resection. Allergy or adverse events related to eradication medication. Administration of proton-pump inhibitor within 2 weeks or Histamine 2 receptor blocker within 1 week.

Administration of these drugs within a week or who need continuous administration of these drugs; aspirin (except low-dose aspirin for primary prophylaxis of cardiovascular disease), intravenous or oral NSAID, anticholinergics, prostaglandin analogs, pro-motility drugs, sucralfate Administration of antibiotics within 4 weeks. Pregnant, breast feeding participant or who do not have a will to avoid pregnancy during clinical trial Administrating one of these drugs (Lovastatin, Simvastatin, Atorvastatin, Indinavir, Ritonavir, Cyclosporin, Terfenadine, Cisapride, Pimozide, Astemizole, HIV protease inhibitors (Atazanavir, Nelfinavir), Ergotamine, Dihydroergotamine, Mizolastine, Bepridil, Ticagrelor) Infectious mononucleosis Central nervous system infection Hematologic disease Galactose intolerance Lactase deficiency Glucose-galactose malabsorption Torsades de pointes.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1230 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | At least 4 weeks from eradication regimen
  Negative urea breath test done

SECONDARY OUTCOMES:
Adverse events | Within one week from eradication administration
  Development of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Wook Kim, MD, PhD, Principal Investigator — Incheon St.Mary's Hospital
Locations (1):
- Incheon St. Mary's Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No